CLINICAL TRIAL: NCT05956678
Title: Implementing and Sustaining a Sleep Treatment to Improve Community Mental Health Part 3: Sustainment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH120147_P3; R01MH120147 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Sleep Wake Disorders; Circadian Rhythm Disorders
Keywords: Implementation; Sustainment; Evidence-based treatment; Community mental health
MeSH Terms: conditions — Sleep Wake Disorders; Chronobiology Disorders | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: CMHC providers are cluster-randomized to either Standard TranS-C or Adapted TranS-C by their CMHC of employment.
Who Masked: Participant
Masking Description: CMHC providers (i.e., the study participants) are blind to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard TranS-C (Experimental): Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
  Interventions: Behavioral: Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)
- Adapted TranS-C (Experimental): The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions and is comprised of 4 cross-cutting interventions featured in every session, 5 modules that apply to the vast majority of patients, and 1 optional module used less commonly, depending on the presentation.
  Interventions: Behavioral: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)

INTERVENTIONS:
Behavioral: Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) — TranS-C is a psychosocial treatment designed to improve sleep and circadian functioning. It is a modular, psychosocial, skills-based approach. In this study, two version of TranS-C will be tested: Standard and Adapted.
  Arms: Standard TranS-C
Behavioral: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) — The Adapted version was derived from Standard TranS-C. It was developed to improve the fit of the treatment with the CMHC context.
  Arms: Adapted TranS-C

SUMMARY:
Research on the sustainment of implemented evidence-based psychological treatments in routine practice settings, such as community mental health centers, is limited. The goal of this study is to test sustainment predictors, mechanisms, and outcomes of the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) in community mental health centers after implementation efforts have ended. CMHC providers have been trained to deliver a "Standard" or "Adapted" version of TranS-C. Researchers will compare these two groups to evaluate differences--and possible mechanisms--with respect to sustainment outcomes.

DETAILED DESCRIPTION:
More research on the sustainment of implemented evidence-based treatments in routine practice settings, such as community mental health centers (CMHCs), is needed. This study is the third and final phase-i.e., the Sustainment Phase-of a cluster-randomized controlled trial and focuses on CMHC providers' sustainment of the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C). The Sustainment Phase seeks to build on the two earlier phases of the trial-the Implementation Phase (NCT04154631) and Train-the-Trainer Phase (NCT05805657)-during which TranS-C was adapted to fit the CMHC context, and ten CMHCs were cluster-randomized to implement Standard TranS-C or Adapted TranS-C via facilitation and train-the-trainer. Data collection for the Sustainment Phase will commence at least three months after implementation efforts in partnering CMHCs have ended. Note that in this study, sustainment is operationalized per Shediac-Rizkallah and Bone's framework (1998) and defined as continued (a) activities, (b) benefits, and (c) capacity of an intervention after implementation efforts have ended.

Aim 1: Report the sustainment outcomes of TranS-C after implementation support has ended.

Aim 2: Evaluate whether manipulating fit to context predicts sustainment outcomes. It is hypothesized that providers in Adapted TranS-C will report better sustainment outcomes (i.e., activities, benefits, and capacity) relative to Standard TranS-C.

Aim 3: Test whether provider perceptions of fit-operationalized as acceptability, appropriateness, and feasibility-mediate the relation between treatment condition (Standard versus Adapted TranS-C) and sustainment outcomes. It is hypothesized that Adapted TranS-C, compared to Standard TranS-C, will predict better sustainment outcomes (i.e., activities, benefits, and capacity) indirectly through better provider perceptions of fit.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for CMHCs are:

* Publicly funded adult mental health outpatient services
* Support from CMHC leadership

The inclusion criteria for CMHC providers are:

* Employed, able to deliver, or have delivered patient-facing services to patients within a CMHC
* Have attended a TranS-C training
* CMHC site of employment has been in a period of sustainment (i.e., implementation activities have ended) for at least three months
* volunteer to participate and formally consent to participate

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Provider Report of Sustainment Scale | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers' continued delivery of TranS-C via three self-report items that are rated on a scale from 0 (not at all) to 4 (to a very great extent) such that higher scores indicate more sustainment.
Adaptations to Evidence-Based Practices Scale | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses provider adaptations to TranS-C via six self-report items that are rated on scale from 1 (not at all) to 4 (very great extent) such that higher scores indicate greater use of adaptations.
Penetration of TranS-C in Provider Caseload | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Two self-report items are used to derive the proportion of eligible patients with whom the provider has used TranS-C (i.e., number of eligible patients with whom provider has used TranS-C / the number of providers' patients with sleep problems), with higher scores indicating more penetration.
Outcomes and Effectiveness Scale | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers' perceptions of TranS-C's health benefits using five self-report items rated on a scale from 0 (to little or no extent) to 7 (to a very great extent) such that higher scores indicate more perceived benefits.
Skills Subscale from the Determinants of Implementation Behavior Questionnaire | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers perceptions of their skills to deliver TranS-C using three self-report items rated on a scale from 1 (strongly disagree) to 7 (strongly agree), where higher scores indicate perceptions of greater skills.
Organizational Resources Subscale from the Implementation Potential Scales | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers' perceptions of whether they have the resources, support, and time needed to deliver TranS-C. Three items are rated on a scale from 1 (strongly disagree) to 6 (strongly agree), where higher ratings indicate more perceived resources, support, and time.

SECONDARY OUTCOMES:
TranS-C Delivery Relative to Pre-Sustainment | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Uses one self-report item to assess whether providers are using TranS-C "more" (scored as 2), "about the same" (scored as 1), or "less" (scored as 0), relative to before the Sustainment Phase.
TranS-C Provider Checklist | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses which TranS-C modules were delivered by providers during the Sustainment Phase using a self-report checklist containing all the modules for each condition. For each module, the checklist is scored such that 0 indicates that the provider did not deliver the module and 1 indicates that the provider delivered the module.
Adaptations Checklist from the Framework for Reporting Adaptations and Modification - Expanded | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses whether providers made any adaptations to TranS-C based on patient characteristics using a self-report checklist. Each patient characteristic on the checklist is scored such that 0 indicates that the provider did not make adaptations based on the characteristic and 1 indicates that the provider did make adaptations based on the characteristic.
Use of Provider Manual and Patient Workbook | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses the extent to which providers follow the TranS-C provider manual and patient workbook via one self-report item with the following scale: 0% (not at all) to 100% (always/completely).
Percentage of TranS-C Strategies Used | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses the percentage of TranS-C strategies used by providers on average when delivering TranS-C to patients via one self-report item with the following scale: 0% (no strategies) to 100% (all the strategies).
TranS-C as Integrated or Standalone Treatment | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses whether providers deliver TranS-C as a standalone intervention using one self-report item with the following 4 categorically-coded response options: I always deliver the sleep treatment as a stand-alone intervention; I sometimes integrate the sleep treatment with other interventions or topics; I always integrate the sleep treatment with other interventions or topics; not applicable.
Number of Sessions with TranS-C | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses the number of sessions in which providers use TranS-C concepts for each patient, on average, via one self-report item that ranges from 0 (no sessions) to 50 (50 sessions).
Creation of Sleep Treatment Materials | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses whether providers have created their own sleep treatment materials via one self-report item with the following categorically-coded response options: no, not relevant, yes with option to describe materials.
Administrator Support Subscale from the Implementation Potential Scales | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses the extent to which providers perceive they have support from leadership and supervisors to deliver TranS-C. Three items are rated on a scale from 1 (strongly disagree) to 6 (strongly agree), where higher scores indicate more support.
Knowledge of TranS-C | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses the extent to which providers (1) understand the theory and concepts behind TranS-C and (2) have the knowledge to conduct TranS-C. Two items are rated on a scale from 0 (not at all) to 7 (extremely), where higher scores indicate more knowledge.

OTHER OUTCOMES:
Acceptability of Intervention Measure | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses provider perceptions of TranS-C's acceptability via four self-report items rated on a scale from 1 (completely disagree) to 5 (completely agree), with higher scores indicating greater acceptability.
Intervention Appropriateness Measure | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses provider perceptions of TranS-C's appropriateness via four self-report items rated on a scale from 1 (completely disagree) to 5 (completely agree), with higher scores indicating greater appropriateness.
Feasibility of Intervention Measure | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses provider perceptions of TranS-C's feasibility via four self-report items rated on a scale from 1 (completely disagree) to 5 (completely agree), with higher scores indicating greater feasibility.
Semi-structured interview with providers | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers' perceptions of TranS-C.
Adaptations in Response to Cultural Backgrounds of Patients | Once during the Sustainment Phase, at least 3 months after implementation efforts have ended.
  Assesses providers' adaptations to TranS-C based on cultural backgrounds of clients. Eight items are rated on a scale from 0 (not at all) to 5 (very great extent), with higher numbers indicating greater use of adaptations.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley; Laurel Sarfan, PhD, Principal Investigator — University of California, Berkeley
Locations (10):
- United States (10):
  - Contra Costa Health, Housing, and Homeless Services Division, Concord, California
  - Solano County Department of Health & Social Services, Behavioral Health Services, Fairfield, California
  - Santa Barbara County Department of Behavioral Wellness, Goleta, California
  - Kings County Behavioral Health, Hanford, California
  - Lake County Behavioral Health Services, Lucerne, California
  - Alameda County Behavioral Health Care Services, Oakland, California
  - Placer County Health and Human Services, Adult System of Care, Roseville, California
  - Monterey County Behavioral Health, Salinas, California
  - Bay Area Community Health, San Jose, California
  - County of Santa Cruz Behavioral Health Services for Children and Adults, Santa Cruz, California

REFERENCES:
- [Derived] Sarfan LD, Agnew ER, Diaz M, Cogan A, Spencer JM, Esteva Hache R, Wiltsey Stirman S, Lewis CC, Kilbourne AM, Harvey AG. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) for serious mental illness in community mental health part 3: study protocol to evaluate sustainment in a hybrid type 2 effectiveness-implementation cluster-randomized trial. Trials. 2024 Jan 15;25(1):54. doi: 10.1186/s13063-023-07900-1. PMID 38225677
- [Derived] Sarfan LD, Agnew ER, Diaz M, Cogan A, Spencer JM, Hache RE, Stirman SW, Lewis CC, Kilbourne AM, Harvey A. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) for serious mental illness in community mental health part 3: Study protocol to evaluate sustainment in a hybrid type 2 effectiveness-implementation cluster-randomized trial. Res Sq [Preprint]. 2023 Oct 30:rs.3.rs-3328993. doi: 10.21203/rs.3.rs-3328993/v1. PMID 37961426